CLINICAL TRIAL: NCT07367243
Title: Acute Effects of Percussive Massage Therapy Applied to Healthy Individuals on Gastrocnemius Muscle Architecture: A Randomized Controlled Trial
Brief Title: Percussive Massage Therapy and Muscle Architecture
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karadeniz Technical University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Murat Emirzeoglu, Assistant Professor, Karadeniz Technical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2025-69
Record Dates: First submitted 2026-01-16; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Muscle Architecture

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Percussive Massage Therapy (PMT) (Experimental): Participants in this arm receive percussive massage therapy applied to the plantar flexor muscle groups of both legs. The intervention is administered for 8 minutes under standardized conditions.
  Interventions: Other: Percussive Massage Therapy (PMT)
- Control Group (No Intervention): Participants in this arm do not receive any intervention and rest in a prone position.

INTERVENTIONS:
Other: Percussive Massage Therapy (PMT) — Percussive massage therapy is applied to the plantar flexor muscle groups of both legs for 8 minutes using standardized procedures.
  Arms: Percussive Massage Therapy (PMT)

SUMMARY:
Percussive massage therapy (PMT) is widely used in therapeutic and athletic settings, but its effects on muscle architecture are not yet fully understood. This study aims to examine the acute effects of PMT applied to the plantar flexor muscles on the muscle architecture of the medial and lateral gastrocnemius muscles in healthy adults aged 18 to 30 years. Participants will be randomly assigned to either a PMT group or a control group. Ultrasonographic assessments will be performed before and after the intervention to evaluate muscle thickness, pennation angle, and fascicle length. The findings of this study may help clarify the acute effects of PMT on muscle structure.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 30 years

Exclusion Criteria:

* History of any surgical procedure
* Hospitalization for any reason within the last two years
* Hospital admission for treatment purposes within the last six months
* Use of any medication within the last three months
* History of congenital, neurological, orthopedic, rheumatologic, or cardiopulmonary pathology or anomaly
* Presence of any known serious systemic disease
* Current health-related complaints or symptoms
* Body mass index (BMI) of 25 kg/m² or higher

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-11-17 (Actual); Primary Completion 2026-02-10 (Estimated); Study Completion 2026-02-10 (Estimated)

PRIMARY OUTCOMES:
Muscle Architecture | Immediately before and immediately after the intervention
  Changes in gastrocnemius medialis and gastrocnemius lateralis muscle architecture, including muscle thickness, pennation angle, and fascicle length, are assessed using ultrasonography.

CONTACTS AND LOCATIONS:
Locations (1):
- Karadeniz Technical University, Trabzon, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No